CLINICAL TRIAL: NCT06403111
Title: Fecal Microbiota Transplantation Combined with Platinum-based Doublet Chemotherapy and Tislelizumab As First-line Treatment for Driver-gene Negative Advanced Non-small-cell Lung Cancer (NSCLC): Study Protocol for a Prospective, Multi-center, Single-arm Exploratory Trial
Brief Title: FMT+Immunotherapy+Chemotherapy As First-line Treatment for Driver-gene Negative Advanced NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Changzhou No.2 People's Hospital (Other)
Responsible Party: Principal Investigator, Hua Jiang, Chief Director of Oncology Department, Changzhou No.2 People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2024]YLJSA005
Record Dates: First submitted 2024-04-27; First posted 2024-05-07 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-08

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chemotherapy+Immunotherapy+FMT (Experimental)
  Interventions: Combination Product: Fecal Microbiota Transplantation (FMT)+chemotherapy+immunotherapy

INTERVENTIONS:
Combination Product: Fecal Microbiota Transplantation (FMT)+chemotherapy+immunotherapy — Participants will receive FMT combined with tislelizumab + pemetrexed + platinum-based treatment (lung adenocarcinoma) / albumin-bound paclitaxel + platinum-based treatment (lung squamous cell carcinoma) for 4-6 cycles. If there is no progression of the disease after 4-6 cycles of the first-line treatment, then patients will enter the maintenance treatment stage. Patients will receive tislelizumab maintenance treatment (lung squamous cell carcinoma), or tislelizumab + pemetrexed maintenance treatment (lung adenocarcinoma).

SUMMARY:
This study plans to reconstruct intestinal microecology through fecal microbiota transplantation (FMT), and combine with standard first-line therapy to enhance the anti-tumor immune effect at the same time, thereby extending the progression-free survival of patients and improving the prognosis of patients.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multi-center, exploratory clinical study. That is, eligible patients with driver-gene negative, ECOG PS 0-1, PD-L1<50% advanced non-small cell lung cancer who have not received prior treatment will be screened after signing informed consent and receive FMT combined with tislelizumab + pemetrexed + platinum-based treatment (lung adenocarcinoma) / albumin-bound paclitaxel + platinum-based treatment (lung squamous cell carcinoma) for 4-6 cycles. If there is no progression of the disease after 4-6 cycles of the first-line treatment, then patients will enter the maintenance treatment stage. Patients will receive tislelizumab maintenance treatment (lung squamous cell carcinoma), or tislelizumab + pemetrexed maintenance treatment (lung adenocarcinoma). RECIST v1.1 was used for tumor evaluation every 6 weeks during treatment. NCI-CTCAE 5.0 was used for safety assessment every 3 weeks. Adverse events were recorded throughout the study to 30 days after the end of treatment. Treatment continues until disease progression, subject withdraws informed consent, loss of follow-up, or death. Patients should provide 10ml whole blood samples and fecal samples at baseline, after two cycles of treatment, before maintenance treatment, and after two cycles of maintenance treatment for the detection of efficacy prediction markers (each cycle is 21 days).

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily joined the study and were able to sign the informed consent with good compliance;
2. Age 18-80 years old (when signing the informed consent form);
3. Patients with histologically or cytologically proven locally advanced (stage IIIB/IIIC), metastatic, or recurrent (stage IV) NSCLC who are inoperable and unable to receive radical concurrent chemoradiotherapy, according to the International Association for the Study of Lung Cancer and the American Joint Committee on Cancer Classification, 8th Edition TNM Classification of Lung cancer;
4. Have not received systemic intravenous anti-tumor therapy before, and the driver gene is negative;
5. PD-L1 expression < 50%;
6. According to the solid tumor efficacy evaluation criteria (RECIST version 1.1), there is at least one radiographically measurable lesion; That is, in CT or MRI detection, the longest diameter of a single lesion was ≥10mm, or the pathological enlargement of a single lymph node was ≥15mm.
7. The physical status score of Eastern Tumor Collaboration Group (ECOG) was 0-1;
8. Expected survival > 3 months;
9. Have adequate organ and bone marrow function, laboratory examination within 7 days prior to enrollment meets the following requirements (no blood components, cell growth factors, albumin or other corrective drugs are allowed within 14 days prior to obtaining laboratory examination), as follows: 1) Blood routine: absolute neutrophil count (ANC) ≥1.5×10 9/L, platelet (PLT) ≥75×10 9/L, hemoglobin (HGB) ≥90 g/L (no blood transfusion or erythropoietin dependence within 14 days); 2) Liver function: serum total bilirubin (TBIL) ≤2 times the upper limit of normal (ULN); Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤ 5x ULN, serum albumin ≥28 g/L; alkaline phosphatase (ALP) ≤5×ULN; 3) Renal function: serum creatinine (Cr) ≤1.5×ULN, or creatinine clearance ≥50 mL/min (using the standard Cockcroft-Gault formula) : Urine routine results showed urinary protein < 2+; For patients with urine protein ≥2+ at baseline, 24-hour urine collection and 24-hour urine protein quantification < 1g should be performed. 4) Coagulation function: International standardized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN; If the subject is receiving anticoagulant therapy, as long as the INR is within the intended range of anticoagulant drug use.
10. For female subjects of reproductive age, a urine or serum pregnancy test should be performed and the result is negative 3 days prior to receiving the initial study drug administration;
11. Subjects and their sexual partners are required to use a medically approved contraceptive method (such as an intrauterine device (IUD), contraceptive pill, or condom) during the study treatment period and for 6 months after the end of the study treatment period.

Exclusion Criteria:

1. Currently participating in an interventional clinical study or receiving another investigational drug or investigational device within 4 weeks prior to initial dosing;
2. Received proprietary Chinese medicines with anti-tumor indications or immunomodulatory drugs (thymosin, interferon, interleukin, etc.) within 2 weeks before the first administration, or received major surgical treatment within 3 weeks before the first administration;
3. Class III - IV congestive heart failure (New York Heart Association classification), poorly controlled and clinically significant arrhythmias;
4. Any arterial thrombosis, embolism or ischemia, such as myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack, occurred within 6 months before treatment;
5. Known allergic reaction to the drug in this study;
6. Patients who require long-term oral, intravenous, or intramuscular administration of systemic corticosteroids;
7. Symptomatic central nervous metastases. Patients with asymptomatic brain metastases (BMS) or BMS whose symptoms are stable after treatment are eligible to participate in this study if they meet all of the following criteria: measurable lesions outside the central nervous system; No midbrain, pontine, cerebellum, meninges, medulla oblongata or spinal cord metastasis; Maintain clinical stability for at least 2 weeks; Stop hormone therapy 3 days before the first dose of the study drug;
8. There is an active infection requiring treatment or systemic anti-infective drugs have been used in the week prior to the first dosing;
9. Has not fully recovered from toxicity and/or complications caused by any intervention before starting treatment (i.e., ≤ grade 1 or baseline, excluding weakness or hair loss);
10. Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive);
11. Untreated active hepatitis B (defined as HBsAg positive and HBV-DNA copy number detected greater than the upper limit of normal value in the laboratory of the study center);
12. Active HCV-infected subjects (HCV antibody positive and HCV-RNA levels above the lower limit of detection);
13. Received live vaccine within 30 days prior to the first dose (cycle 1, day 1); Note: Injectable inactivated virus vaccine against seasonal influenza is permitted for 30 days prior to initial administration; However, live attenuated influenza vaccines administered intranasally are not permitted.
14. Pregnant or lactating women;
15. Medical history or evidence of disease that may interfere with test results, prevent participants from fully participating in the study, abnormal treatment or laboratory test values, or other conditions that the investigator considers unsuitable for enrollment The Investigator considers other potential risks unsuitable for participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
12-Months Progression-Free Survival Rate (12month-PFS) | up to 12 months
  The proportion of patients whose disease did not progress 12 months after treatment

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 12 months
  Objective response rate will be assessed by investigators.
Median Progression-Free Survival (mPFS) | up to 12 months
  Observation for mPFS will be recorded until the end of follow-up after the start of 1st cycle of treatment.
Incidence of Adverse events (AEs) | up to 12 months
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).
Duration of Response (DOR) | up to 12 months
  The time between the first assessment of a tumor as CR or PR and the first assessment as progressive disease (PD) or death from any cause.
The Diversity of Fecal Microbiota | up to 12 months
  This will be detected by 16s rRNA sequencing or metagenomes.
Quality of Life (QoL) | up to 12 months
  QoL will be evaluated by EORTC-QLQ-C30.

CONTACTS AND LOCATIONS:
Overall Officials: Hua Jiang, MD, Study Director — Changzhou No.2 People's Hospital
Locations (1):
- Changzhou No.2 Poeple's Hospital, Changzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wei Y, Qin L, Wu X, Li D, Qian D, Jiang H, Geng Q. Faecal microbiota transplantation combined with platinum-based doublet chemotherapy and tislelizumab as first-line treatment for driver-gene negative advanced non-small cell lung cancer (NSCLC): study protocol for a prospective, multicentre, single-arm exploratory trial. BMJ Open. 2025 Mar 4;15(3):e094366. doi: 10.1136/bmjopen-2024-094366. PMID 40037667